CLINICAL TRIAL: NCT05189249
Title: Determinant of Repeat Revascularization Within 5 Years of Percutaneous Coronary Intervention at a Tertiary Care Hospital, Karachi: A Matched Case-Control Study
Brief Title: Determinant of Repeat Revascularization After Percutaneous Coronary Intervention
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Komal Valliani, Principal Investigator, Aga Khan University
Other Study IDs: 5004-CHS-ERC-17
Record Dates: First submitted 2021-12-28; First posted 2022-01-12 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Percutaneous Coronary Intervention; Coronary Artery Disease
Keywords: Repeat revascularization; Percutaneous Coronary Intervention; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Patients who have undergone repeat revascularization within 5 years of undergoing index PCI at Aga Khan University Hospital Karachi.
  Interventions: Other: No intervention performed
- Control: Patients who have not undergone repeat revascularization within 5 years of undergoing index PCI at Aga Khan University Hospital Karachi.
  Interventions: Other: No intervention performed

INTERVENTIONS:
Other: No intervention performed — No intervention performed. Participants were enrolled retrospectively and medical records were accessed for data.

SUMMARY:
To determine factors associated with repeat revascularization among adults aged 25 years and above within 5 years of first Percutaneous Coronary Intervention (PCI) at a tertiary care hospital.

DETAILED DESCRIPTION:
Matched case-control study design was employed to determine the association between re-peat revascularization and its determinants in patients within 5 years of undergoing index PCI. The case was defined as a patient who had undergone repeat revascularization within 5 years of undergoing index PCI. Control was defined as a patient who had not undergone repeat revascularization within 5 years of undergoing index PCI.

The retrospective study was carried out with the approval of the Ethical Review Committee of the tertiary care hospital where the study was carried out. A waiver of informed consent was granted as this was a retrospective study and all patients were discharged from the hospital.

A minimum of 120 cases with matched 240 controls were required in 1:2 case to control ratio. This sample size was essential to achieve the power of 80% for an anticipated matched odds ratio of 2 with the hypothesized correlation of 0.2 using a two-sided hypothesis test with a significance level of 0.05.

The outcome of the study was the Repeat revascularization status. There are different types of repeat revascularization according to the site and lesion to which intervention has been provided. Any type of repeat revascularization was considered and enrolled as a case in this study5.

Covariates included in the study were divided into patient characteristics (gender, age, health coverage, BMI, smoking status), comorbidity status (Hypertension, Diabetes Mellitus, Hyperlipidaemia, valvular disease), clinical characteristics (Creatinine level, Systolic Blood Pressure, Diastolic Blood Pressure, HbA1c, Cholesterol level, other technical factors related to the index PCI) and medication status (Beta-blocker, ACE Inhibitor, Statin).

ELIGIBILITY:
Inclusion Criteria for Cases:

* Aged 25 years and older
* Undergone repeat revascularization within 5 years of undergoing index PCI (from 2011 to 2017).

Exclusion Criteria for Cases:

* If suffering from any hypercoagulable disorder
* Revascularization procedure was per-formed outside the study setting
* Staged PCI within 3 weeks or planned PCI within 6 months of Index PCI.

Inclusion Criteria for Controls:

* Patients aged 25 years and older
* Undergone PCI once from the year 2011 to 2017.

Exclusion Criteria for Controls:

* If suffering from any hypercoagulable disorder.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population includes all the adult patients age 25 years and above who were revascularized at least at the Aga Khan University Hospital, Karachi.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Factors associated with repeat revascularization | January 2018 to December 2018
  Identify factors that are associated with repeat coronary intervention in the form of PCI or CABG once patient has been discharged after index PCI and during follow-up years (excluding staged PCI planned within three weeks of index PCI).

CONTACTS AND LOCATIONS:
Overall Officials: Komal Valliani, BScN, MScEB, Principal Investigator — Aga Khan University Karachi
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan